CLINICAL TRIAL: NCT06070649
Title: The Potential Therapeutic Effects of Psychedelic, N, N-dimethyltryptamine (DMT), on Alcohol Use Disorder (AUD)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Anahita Bassir Nia, Assistant Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2000035937; 1R21AA030649-01A1 (NIH)
Record Dates: First submitted 2023-08-16; First posted 2023-10-06 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Alcohol Use Disorder (AUD); Alcohol-Related Disorders; Alcohol Use
MeSH Terms: conditions — Alcoholism; Alcohol-Related Disorders; Alcohol Drinking | interventions — N,N-Dimethyltryptamine; Diphenhydramine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator): Bolus of 0.3mg/kg/min DMT (5min) + Normal Saline infusion (60 min)
  Interventions: Drug: 0.3mg/kg/min Dimethyltryptamine + Normal Saline infusion
- Group 2 (Active Comparator): Bolus of 0.2 mg/kg/min DMT (5 min) + 0.01mg/kg/min infusion (60 min)
  Interventions: Drug: 0.2 mg/kg/min + Dimethyltryptamine 0.01mg/kg/min infusion
- Group 3 (Placebo Comparator): Bolus of 25 mg Diphenhydramine (5 min) + Normal Saline infusion (60 min)
  Interventions: Drug: 25 mg Diphenhydramine (5 min) + Normal Saline

INTERVENTIONS:
Drug: 0.3mg/kg/min Dimethyltryptamine + Normal Saline infusion — Infusion
  Other Names: Moderate Dose DMT
  Arms: Group 1
Drug: 0.2 mg/kg/min + Dimethyltryptamine 0.01mg/kg/min infusion — Infusion
  Other Names: Low Dose DMT
  Arms: Group 2
Drug: 25 mg Diphenhydramine (5 min) + Normal Saline — Infusion
  Arms: Group 3

SUMMARY:
This proposed study is a double-blind, randomized, placebo-controlled, parallel-group, laboratory study to determine the effects of DMT, plus psychotherapy, on Alcohol Use Disorder.

DETAILED DESCRIPTION:
This study is a placebo-controlled, randomized, double blind, clinical trial to investigate the safety, tolerability and efficacy of the psychedelic dimethyltryptamine (DMT), in addition to a short course of psychotherapy, on Alcohol Use Disorder (AUD). The investigators hypothesize that relative to control (0.2 mg/kg/min + Dimethyltryptamine 0.01mg/kg/min infusion plus psychotherapy), a single psychedelic dose of DMT (plus psychotherapy) in individuals with AUD will 1) be safe and 2) well-tolerated, and 3) reduce alcohol consumption measured in the laboratory the day after, and over the following 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual of Mental Disorders-5th edition (DSM-5) diagnosis of Alcohol Use Disorder
* Medically healthy
* Ability to provide consent

Exclusion Criteria:

* Unstable medical conditions

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of DMT in women and men with AUD | Day 0 through Day 56
  Systematic Assessment for Treatment Emergent Effects (SAFTEE) and MedDRA will be used weekly for 8 weeks to assess safety and tolerability of DMT in women and men with AUD.
The effects of DMT, plus psychotherapy, on alcohol consumption | Day 0 through Day 56
  We will assess the desire of participants to drink alcohol in an experimental setting using the Alcohol Drinking Paradigm.

SECONDARY OUTCOMES:
The relationship between acute psychedelic effects of DMT and alcohol consumption | Day 0 through Day 56
  The Mystical Experience Questionnaire (MEQ) will be used to assess the relationship between acute psychedelic effects of DMT and alcohol consumption.
The relationship between acute psychedelic effects of DMT and alcohol consumption | Day 0 through Day 56
  The Ego-Dissolution Inventory (EDI) will be used to assess the relationship between acute psychedelic effects of DMT and alcohol consumption.
The long-term effects of a single dose of DMT, plus psychotherapy, on alcohol consumption over the subsequent 8 weeks. | Day 0 through Day 56
  The Timeline Followback (TLFB) approach will be used to assess the long-term effects of a single dose of DMT, plus psychotherapy on alcohol consumption.
The long-term effects of a single dose of DMT, plus psychotherapy, on alcohol consumption over the subsequent 8 weeks. | Day 0 through Day 56
  Stages of Change Readiness and Treatment Eagerness Scale (SOCRATES) will be used to assess the long-term effects of a single dose of DMT, plus psychotherapy on alcohol consumption.
The long-term effects of a single dose of DMT, plus psychotherapy, on alcohol consumption over the subsequent 8 weeks. | Day 0 through Day 56
  Substance use disorder behaviors and risks with the Brief Addiction Monitor (BAM) will be used to assess the long-term effects of a single dose of DMT, plus psychotherapy on alcohol consumption.
The prosocial effects of DMT, plus psychotherapy, and changes in personality traits | Day 0 through Day 56
  Prosocial effects with be assessed using the Prosocial Personality Battery (PSP). The scale consists of 56 total items and uses a Likert-type scale with 5 answer-choices.
The prosocial effects of DMT, plus psychotherapy, and changes in personality traits | Day 0 through Day 56
  Prosocial effects with be assessed using the Social Connectedness Scale - Revised (SCS-R).
The prosocial effects of DMT, plus psychotherapy, and changes in personality traits | Day 0 through Day 56
  Prosocial effects with be assessed using the Mindful Attention Awareness Scale (MAAS).
The relationship between the intensity of subjective psychedelic experience with lifetime history of chronic stress and trauma | Day 0 through Day 56
  The Life Events Checklist (LEC) will be used to assess the relationship between the intensity of subjective psychedelic experience with lifetime history of chronic stress and trauma.
The relationship between the intensity of subjective psychedelic experience with lifetime history of chronic stress and trauma | Day 0 through Day 56
  The Childhood Trauma Questionnaire (CTQ-SF) will be used to assess the relationship between the intensity of subjective psychedelic experience with lifetime history of chronic stress and trauma.

CONTACTS AND LOCATIONS:
Overall Officials: Anahita Bassir Nia, MD, Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States